CLINICAL TRIAL: NCT03601637
Title: A Phase 3, 2-part, Open-label Study to Evaluate the Safety and Pharmacokinetics of Lumacaftor/Ivacaftor in Subjects 1 to Less Than 2 Years of Age With Cystic Fibrosis, Homozygous for F508del
Brief Title: Safety and Pharmacokinetic Study of Lumacaftor/Ivacaftor in Participants 1 to Less Than 2 Years of Age With Cystic Fibrosis, Homozygous for F508del
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VX16-809-122; 2017-004794-13 (EudraCT Number)
Record Dates: First submitted 2018-07-18; First posted 2018-07-26 (Actual); Results first posted 2023-01-06 (Actual); Last update posted 2023-01-06 (Actual); Status verified 2022-12

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — lumacaftor; ivacaftor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part A: LUM/IVA (Experimental): Participants weighing 7 to less than (<)10 kilograms (kg) at screening received LUM 75 milligrams (mg)/IVA 94 mg fixed-dose combination (FDC) every 12 hours (q12h) and those weighing 10 to <14 kg at screening received LUM 100 mg/IVA 125 mg q12h for 15 days. Participants weighing greater than or equal to (>=)14 kg at screening received LUM 150 mg/IVA 188 mg FDC q12h for 15 days.
  Interventions: Drug: LUM; Drug: IVA
- Part B: LUM/IVA (Experimental): Participants weighing 7 to <9 kg at screening received LUM 75 mg/IVA 94 mg FDC q12h and those weighing 9 to <14 kg received LUM 100 mg/IVA 125 mg q12h for 24 weeks. Participants weighing >=14 kg at screening received LUM 150 mg/IVA 188 mg FDC q12h for 24 weeks. Doses were adjusted upwards for changes in weight.
  Interventions: Drug: LUM; Drug: IVA

INTERVENTIONS:
Drug: LUM — Fixed Dose Combination (FDC) granules (LUM/IVA).
  Other Names: lumacaftor; VX-809
Drug: IVA — FDC granules (LUM/IVA).
  Other Names: ivacaftor; VX-770

SUMMARY:
This study will evaluate the safety and pharmacokinetics (PK) of lumacaftor (LUM) and ivacaftor (IVA) in participants 1 to less than 2 years of age with cystic fibrosis (CF), homozygous for F508del (F/F).

ELIGIBILITY:
Key Inclusion Criteria:

* Participants will be 1 to less than 2 years of age on day 1 of the relevant part of the study
* Homozygous for F508del (F/F)

Key Exclusion Criteria:

* Any clinically significant laboratory abnormalities at the screening visit that would interfere with the study assessments or pose an undue risk for the participants
* Solid organ or hematological transplantation

Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 12 Months to 23 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 61 (Actual)
Dates: Start 2018-09-07 (Actual); Primary Completion 2021-10-29 (Actual); Study Completion 2021-10-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (27):
- United States (24):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Stanford University, Palo Alto, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Yale New Haven Medical Center, New Haven, Connecticut
  - Nemours / Alfred I. duPont Hospital for Children, Wilmington, Delaware
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Ann & Robert Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Riley Hospital for Children at Indiana University Health, Indianapolis, Indiana
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - Children's Respiratory and Critical Care Specialists, P.A., Children's Hospitals and Clinics of Minnesota, Minneapolis, Minnesota
  - The Children's Mercy Hospital, Kansas City, Missouri
  - Cardinal Glennon Children's Hospital - St. Louis University, St Louis, Missouri
  - University of Rochester Medical Center, Rochester, New York
  - University of North Carolina Hospitals, Chapel Hill, North Carolina
  - Wake Forest University School of Medicine - Brenner Children's Hospital, Winston-Salem, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Medical Center of Dallas, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - University of Utah / Primary Children's Medical Center, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
- Canada (3):
  - McGill University Health Centre, Glen Site, Montreal Children's Hospital, Montreal
  - The Hospital for Sick Children, Toronto
  - British Columbia's Children's Hospital, Vancouver

IPD SHARING:
Plan to Share IPD: No
Details on Vertex data sharing criteria and process for requesting access can be found at: https://www.vrtx.com/independent-research/clinical-trial-data-sharing

REFERENCES:
- [Derived] Heneghan M, Southern KW, Murphy J, Sinha IP, Nevitt SJ. Corrector therapies (with or without potentiators) for people with cystic fibrosis with class II CFTR gene variants (most commonly F508del). Cochrane Database Syst Rev. 2023 Nov 20;11(11):CD010966. doi: 10.1002/14651858.CD010966.pub4. PMID 37983082
- [Derived] Rayment JH, Asfour F, Rosenfeld M, Higgins M, Liu L, Mascia M, Paz-Diaz H, Tian S, Zahigian R, McColley SA. A Phase 3, Open-Label Study of Lumacaftor/Ivacaftor in Children 1 to Less Than 2 Years of Age with Cystic Fibrosis Homozygous for F508del-CFTR. Am J Respir Crit Care Med. 2022 Nov 15;206(10):1239-1247. doi: 10.1164/rccm.202204-0734OC. PMID 35771568
- [Derived] Southern KW, Murphy J, Sinha IP, Nevitt SJ. Corrector therapies (with or without potentiators) for people with cystic fibrosis with class II CFTR gene variants (most commonly F508del). Cochrane Database Syst Rev. 2020 Dec 17;12(12):CD010966. doi: 10.1002/14651858.CD010966.pub3. PMID 33331662

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study was conducted in participants with cystic fibrosis (CF) aged 1 through less than 2 years of age who are homozygous for F508del. A total of 61 participants were enrolled in Parts A and B of the study. One participant in Part B was enrolled but not dosed in this study. Therefore, data for 60 participants are reported in the participant flow and baseline characteristics sections.
Groups:
- Part A: LUM/IVA: Participants weighing 7 to less than( <)10 kilograms (kg) at screening received lumacaftor (LUM) 75 milligrams (mg)/ ivacaftor (IVA) 94 mg fixed-dose combination (FDC) every 12 hours (q12h) and those weighing 10 to <14 kg at screening received LUM 100 mg/IVA 125 mg q12h for 15 days. Participants weighing greater than or equal to (>=)14 kg at screening received LUM 150 mg/IVA 188 mg FDC q12h for 15 days.
Period: Overall Study
Arm/Group | Part A: LUM/IVA | Part B: LUM/IVA
Started | 14 | 46
Completed | 13 | 43
Not Completed | 1 | 3
Not completed — Withdrawal of Consent (not due to adverse event) | 0 | 1
Not completed — Adverse Event | 1 | 1
Not completed — Other | 0 | 1

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of the study drug during the treatment period were included in the baseline analysis. The baseline analysis was collected for the overall treatment arm, irrespective of a weight-based dose regimen. Therefore, the analysis is reported in a single arm for each study part (Part A: LUM/IVA and Part B: LUM/IVA).
Groups:
- Part A: LUM/IVA: Participants weighing 7 to less than(<)10 kilograms (kg) at screening received lumacaftor (LUM) 75 milligrams (mg)/ ivacaftor (IVA) 94 mg fixed-dose combination (FDC) every 12 hours (q12h) and those weighing 10 to <14 kg at screening received LUM 100 mg/IVA 125 mg q12h for 15 days. Participants weighing greater than or equal to (>=)14 kg at screening received LUM 150 mg/IVA 188 mg FDC q12h for 15 days.
- Part B: LUM/IVA: Participants weighing 7 to <9 kg at screening received LUM 75 mg/ IVA 94 mg FDC q12h and those weighing 9 to <14 kg received LUM 100 mg/IVA 125 mg q12h for 24 weeks. Participants weighing >=14 kg at screening received LUM 150 mg/IVA 188 mg FDC q12h for 24 weeks. Doses were adjusted upwards for changes in weight.
- Total: Total of all reporting groups
Arm/Group | Part A: LUM/IVA | Part B: LUM/IVA | Total
Number analyzed (Participants) | 14 | 46 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 14 | 46 | 60
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 24 | 31
  Male | 7 | 22 | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 13 | 37 | 50
  Unknown or Not Reported | 0 | 7 | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 14 | 34 | 48
  Black or African American | 0 | 1 | 1
  Asian | 0 | 0 | 0
  American Indian or Alaska Native | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Not collected per local regulations | 0 | 7 | 7
  Other | 0 | 3 | 3

OUTCOME MEASURES:

1. Primary Outcome: Part A: Observed Plasma Concentrations From 3-4 Hours (C3-4hr) of LUM and IVA
Time Frame: Day 1 and Day 15
Population: Pharmacokinetic (PK) set included participants who received at least 1 dose of study drug. Here the "Number Analyzed" signifies those participants who were evaluable at specified time point.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Groups:
- Part A: LUM 75 mg/IVA 94 mg: Participants received LUM 75 mg /IVA 94 mg dose every 12 hours for 15 days.
- Part A: LUM 100 mg/IVA 125 mg: Participants received LUM 100 mg/IVA 125 mg dose 2 every 12 hours for 15 days.
Arm/Group | Part A: LUM 75 mg/IVA 94 mg | Part A: LUM 100 mg/IVA 125 mg
Number analyzed (Participants) | 7 | 7
nanograms per milliliter (ng/mL)
  Day 1: LUM | 14600 (5560) | 12600 (7190)
  Day 15: LUM: number analyzed (Participants) | 7 | 5
  Day 15: LUM | 16600 (9590) | 13900 (5800)
  Day 1: IVA | 1620 (648) | 1320 (804)
  Day 15: IVA: number analyzed (Participants) | 7 | 5
  Day 15: IVA | 718 (352) | 496 (268)

2. Primary Outcome: Part A: Observed Pre-dose Plasma Concentration (Ctrough) of LUM and IVA
Time Frame: Pre-dose at Day 8 and Day 15
Population: PK set included participants who received at least 1 dose of study drug. Here the "Number Analyzed" signifies those participants who were evaluable at specified time point.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Part A: LUM 75 mg/IVA 94 mg: Participants received LUM 75 mg/IVA 94 mg dose every 12 hours for 15 days.
- Part A: LUM 100 mg/IVA 125 mg: Participants received LUM 100 mg/IVA125 mg dose every 12 hours for 15 days.
Arm/Group | Part A: LUM 75 mg/IVA 94 mg | Part A: LUM 100 mg/IVA 125 mg
Number analyzed (Participants) | 7 | 7
ng/mL
  Day 8: LUM: number analyzed (Participants) | 7 | 6
  Day 8: LUM | 12000 (8880) | 12800 (3900)
  Day 15: LUM: number analyzed (Participants) | 5 | 6
  Day 15: LUM | 8380 (7790) | 10500 (3070)
  Day 8: IVA: number analyzed (Participants) | 7 | 6
  Day 8: IVA | 169 (75.5) | 185 (101)
  Day 15: IVA: number analyzed (Participants) | 5 | 6
  Day 15: IVA | 78.9 (19.1) | 120 (60.5)

3. Primary Outcome: Part B : Safety and Tolerability as Assessed by Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Time Frame: From Day 1 up to Week 26
Population: Safety set included all participants who received at least 1 dose of study drug in the treatment period. The safety and tolerability analyses were assessed for the overall treatment arm, irrespective of weight-based dose regimen. Therefore, the analysis is reported in a single Part B: LUM/IVA arm.
Measure: Number; unit: participants
Groups:
- Part B: LUM/IVA: Participants weighing 7 to <9 kg at screening received LUM 75 mg/IVA 94 mg FDC q12h and those weighing 9 to <14 kg received LUM 100 mg/IVA 125 mg FDC q12h for 24 weeks. Participants weighing >=14 kg at screening received LUM 150 mg/IVA 188 mg FDC q12h for 24 weeks. Doses were adjusted upwards for changes in weight.
Arm/Group | Part B: LUM/IVA
Number analyzed (Participants) | 46
participants
  Participants with TEAEs | 44
  Participants with SAEs | 5

4. Secondary Outcome: Part A: Safety and Tolerability as Assessed by Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Time Frame: From Day 1 up to Day 25
Population: Safety set included all participants who received at least 1 dose of study drug in the treatment period. The safety and tolerability analyses were assessed for the overall treatment arm, irrespective of weight-based dose regimen. Therefore, the analysis is reported in a single Part A: LUM/IVA arm.
Measure: Number; unit: participants
Groups:
- Part A: LUM/IVA: Participants weighing 7 to <10 kg at screening received LUM 75 mg/IVA 94 mg FDC q12h and those weighing 10 to <14 kg at screening received LUM 100 mg/IVA 125 mg FDC q12h for 15 days. Participants weighing >=14 kg at screening received LUM 150 mg/IVA 188 mg FDC q12h for 15 days.
Arm/Group | Part A: LUM/IVA
Number analyzed (Participants) | 14
participants
  Participants with TEAEs | 12
  Participants with SAEs | 0

5. Secondary Outcome: Part A: Observed Pre-dose Plasma Concentration (Ctrough) of LUM and IVA and Their Respective Metabolites (M28-LUM, M1-IVA and M6-IVA)
Time Frame: Pre-dose at Day 8 and Day 15
Population: PK set included participants who received at least 1 dose of study drug. Here the "Number Analyzed signifies those participants who were evaluable at specified time point.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part A: LUM 75 mg/IVA 94 mg | Part A: LUM 100 mg/IVA 125 mg
Number analyzed (Participants) | 7 | 7
ng/mL
  Day 8: M28-LUM: number analyzed (Participants) | 7 | 6
  Day 8: M28-LUM | 1410 (791) | 1470 (365)
  Day 15: M28-LUM: number analyzed (Participants) | 5 | 6
  Day 15: M28-LUM | 1460 (1060) | 1370 (468)
  Day 8: M1-IVA: number analyzed (Participants) | 7 | 6
  Day 8: M1-IVA | 606 (298) | 842 (527)
  Day 15: M1-IVA: number analyzed (Participants) | 5 | 6
  Day 15: M1-IVA | 284 (70.2) | 604 (394)
  Day 8: M6-IVA: number analyzed (Participants) | 7 | 6
  Day 8: M6-IVA | 2380 (843) | 3290 (1830)
  Day 15: M6-IVA: number analyzed (Participants) | 5 | 6
  Day 15: M6-IVA | 1460 (763) | 2800 (2300)

6. Secondary Outcome: Part B: Absolute Change in Sweat Chloride
Time Frame: From Baseline at Week 24
Population: The Full Analysis Set (FAS) included all enrolled participants who were exposed to any amount of study drug in Part B.The pharmacodynamic analyses were assessed for the overall treatment arm, irrespective of weight-based dose regimen. Therefore, the analysis is reported in a single Part B: LUM/IVA arm.
Measure: Mean (Standard Deviation); unit: Millimole per liter (mmol/L)
Arm/Group | Part B: LUM/IVA
Number analyzed (Participants) | 46
Millimole per liter (mmol/L) | -29.1 (13.5)

7. Secondary Outcome: Part B: Observed Pre-dose Plasma Concentration (Ctrough) of LUM and IVA and Their Respective Metabolites (M28-LUM, M1-IVA and M6-IVA)
Time Frame: Pre-dose at Day 15, Week 4, Week 12 and Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Part B: LUM 75 mg/IVA 94 mg: Participants received LUM 75 mg/IVA 94 mg dose every 12 hours for 24 weeks.
- Part B: LUM 100 mg/IVA 125 mg: Participants received LUM 100 mg/IVA 125 mg dose every 12 hours for 24 weeks.
- Part B: LUM 150 mg/IVA 188 mg: Participants received LUM 150 mg/IVA 188 mg dose every 12 hours for 24 weeks.
Arm/Group | Part B: LUM 75 mg/IVA 94 mg | Part B: LUM 100 mg/IVA 125 mg | Part B: LUM 150 mg/IVA 188 mg
Number analyzed (Participants) | 1 | 44 | 1
ng/mL
  Day 15: LUM: number analyzed (Participants) | 1 | 43 | 1
  Day 15: LUM | 13500 | 9030 (4390) | 887
  Week 4: LUM: number analyzed (Participants) | 1 | 43 | 1
  Week 4: LUM | 21900 | 9370 (5030) | 1000
  Week 12: LUM: number analyzed (Participants) | 1 | 41 | 1
  Week 12: LUM | 12100 | 9160 (4400) | 566
  Week 24: LUM: number analyzed (Participants) | 1 | 35 | 1
  Week 24: LUM | 11200 | 8930 (5310) | 288
  Day 15: M28-LUM: number analyzed (Participants) | 1 | 43 | 1
  Day 15: M28-LUM | 1460 | 1260 (528) | 786
  Week 4: M28-LUM: number analyzed (Participants) | 1 | 43 | 1
  Week 4: M28-LUM | 1570 | 1340 (579) | 602
  Week 12: M28-LUM: number analyzed (Participants) | 1 | 41 | 1
  Week 12: M28-LUM | 1740 | 1440 (599) | 501
  Week 24: M28-LUM: number analyzed (Participants) | 1 | 35 | 1
  Week 24: M28-LUM | 1870 | 1470 (548) | 569
  Day 15: IVA: number analyzed (Participants) | 1 | 43 | 1
  Day 15: IVA | 213 | 112 (68.3) | 3.68
  Week 4: IVA: number analyzed (Participants) | 1 | 43 | 1
  Week 4: IVA | 267 | 112 (82.9) | 11.4
  Week 12: IVA: number analyzed (Participants) | 1 | 41 | 1
  Week 12: IVA | 286 | 91.7 (44.7) | 2.18
  Week 24: IVA: number analyzed (Participants) | 1 | 34 | 1
  Week 24: IVA | 37.1 | 144 (296) | 2.86
  Day 15: M1-IVA: number analyzed (Participants) | 1 | 43 | 1
  Day 15: M1-IVA | 1420 | 437 (291) | 18.1
  Week 4: M1-IVA: number analyzed (Participants) | 1 | 43 | 1
  Week 4: M1-IVA | 1930 | 466 (359) | 58.0
  Week 12: M1-IVA: number analyzed (Participants) | 1 | 41 | 1
  Week 12: M1-IVA | 759 | 418 (236) | 18.3
  Week 24: M1-IVA: number analyzed (Participants) | 1 | 35 | 1
  Week 24: M1-IVA | 256 | 499 (613) | 18.5
  Day 15: M6-IVA: number analyzed (Participants) | 1 | 43 | 1
  Day 15: M6-IVA | 4740 | 1930 (1460) | 43.9
  Week 4: M6-IVA: number analyzed (Participants) | 1 | 43 | 1
  Week 4: M6-IVA | 9090 | 1970 (1490) | 131
  Week 12: M6-IVA: number analyzed (Participants) | 1 | 41 | 1
  Week 12: M6-IVA | 3520 | 1950 (1430) | 46.5
  Week 24: M6-IVA: number analyzed (Participants) | 1 | 35 | 1
  Week 24: M6-IVA | 1320 | 1740 (1130) | 63.3

ADVERSE EVENTS:
Time Frame: From Day 1 Through Safety Follow-up Period (up to Day 25 for Part A and up to Week 26 for Part B)
Description: The safety and tolerability analyses were assessed for the overall treatment arm, irrespective of weight-based dose regimen. Therefore, the analysis is reported in a single arm for each study part (Part A: LUM/IVA and Part B: LUM/IVA).
Groups:
- Part A: LUM/IVA: Participants weighing 7 to <10 kg at screening received LUM 75 mg/IVA 94 mg FDC q12h and those weighing 10 to <14 kg at screening received LUM 100 mg/IVA 125 mg q12h for 15 days. Participants >=14 kg at screening received LUM 150 mg/IVA 188 mg FDC q12h for 15 days.
- Part B: LUM/IVA: Participants weighing 7 to <9 kg at screening received LUM 75 mg/ IVA 94 mg FDC q12h and those weighing 9 to <14 kg received LUM 100 mg/IVA 125 mg FDC q12h for 24 weeks. Participants weighing >=14 kg at screening received LUM 150 mg/IVA 188 mg FDC q12h for 24 weeks. Doses were adjusted upwards for changes in weight.
Arm/Group | Part A: LUM/IVA | Part B: LUM/IVA
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/46
Serious Adverse Events (participants affected / at risk) | 0/14 | 5/46
Other Adverse Events (participants affected / at risk) | 12/14 | 42/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: LUM/IVA (N=14) | Part B: LUM/IVA (N=46)
Post procedural fever (Injury, poisoning and procedural complications) | 0 | 1
Distal intestinal obstruction syndrome (Gastrointestinal disorders) | 0 | 1
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 0 | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: LUM/IVA (N=14) | Part B: LUM/IVA (N=46)
Lip injury (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 4
Pseudomonas test positive (Investigations) | 0 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 16
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 5 | 5
Crying (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 10
Insomnia (Psychiatric disorders) | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 3
Constipation (Gastrointestinal disorders) | 1 | 5
Diarrhoea (Gastrointestinal disorders) | 0 | 3
Flatulence (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 8
Rash (Skin and subcutaneous tissue disorders) | 3 | 4
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1
Ear infection (Infections and infestations) | 0 | 5
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 0 | 8
Influenza (Infections and infestations) | 2 | 0
Nasopharyngitis (Infections and infestations) | 0 | 4
Viral upper respiratory tract infection (Infections and infestations) | 0 | 5
Upper respiratory tract infection (Infections and infestations) | 1 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-07-29): https://cdn.clinicaltrials.gov/large-docs/37/NCT03601637/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-19): https://cdn.clinicaltrials.gov/large-docs/37/NCT03601637/SAP_001.pdf